CLINICAL TRIAL: NCT00078117
Title: Suboxone: (Buprenorphine/Naloxone) Comparison of Two Taper Schedules
Brief Title: Suboxone: (Buprenorphine/Naloxone) Comparison of Two Taper Schedules - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Walter Ling, M.D., University of California, Los Angeles
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-CTN-0003-1
Record Dates: First submitted 2004-02-19; First posted 2004-02-20 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2010-04

CONDITIONS: Opioid-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this protocol is to to compare the clinical utility of two dosage tapering regimens in Buprenorphine/Naloxone stabilized subjects for opiate detoxification.

ELIGIBILITY:
Inclusion Criteria:

* Females are not pregnant or lactating
* Subjects meet DSM-IV criteria for opiate dependence, are medically and psychiatrically stable, and do not have a current history of benzodiazepine dependence abuse, dependence, or treatment

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 516
Dates: Start 2003-06; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Opiate abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — University of California, Los Angeles
Locations (11):
- United States (11):
  - Addiction Research & Treatment Services (ARTS), Denver, Colorado
  - Denver Health & Hospitals Authority, Denver, Colorado
  - Hartford Dispensary, Hartford, Connecticut
  - Connecticut Counseling Centers, Waterbury, Connecticut
  - LI Jewish Health System, Glen Oaks, New York
  - New York VA Medical Center, New York, New York
  - South Light-Wakeview Clinic, Raleigh, North Carolina
  - Coastal Horizons Center, Inc., Wilmington, North Carolina
  - CODA, Portland, Oregon
  - Norfolk CSB, Norfolk, Virginia
  - Providence Behavioral Health Services, Everett, Washington

REFERENCES:
- [Derived] Nielsen S, Hillhouse M, Thomas C, Hasson A, Ling W. A comparison of buprenorphine taper outcomes between prescription opioid and heroin users. J Addict Med. 2013 Jan-Feb;7(1):33-8. doi: 10.1097/ADM.0b013e318277e92e. PMID 23222095
- [Derived] Hillhouse M, Canamar CP, Ling W. Predictors of outcome after short-term stabilization with buprenorphine. J Subst Abuse Treat. 2013 Mar;44(3):336-42. doi: 10.1016/j.jsat.2012.08.016. Epub 2012 Sep 26. PMID 23021099
- [Derived] Back SE, Payne RL, Wahlquist AH, Carter RE, Stroud Z, Haynes L, Hillhouse M, Brady KT, Ling W. Comparative profiles of men and women with opioid dependence: results from a national multisite effectiveness trial. Am J Drug Alcohol Abuse. 2011 Sep;37(5):313-23. doi: 10.3109/00952990.2011.596982. PMID 21854273
- [Derived] Ling W, Hillhouse M, Domier C, Doraimani G, Hunter J, Thomas C, Jenkins J, Hasson A, Annon J, Saxon A, Selzer J, Boverman J, Bilangi R. Buprenorphine tapering schedule and illicit opioid use. Addiction. 2009 Feb;104(2):256-65. doi: 10.1111/j.1360-0443.2008.02455.x. PMID 19149822